CLINICAL TRIAL: NCT06784518
Title: Stroke Cerebral Reorganization Pathways Longitudinal Study After Stroke of the Clinical Motor Pattern and the Cerebral Reorganization According to the Different Damaged Motor Pathways (main and Accessory) (SPECTRE)
Brief Title: Stroke Cerebral Reorganization Pathways (SPECTRE)
Acronym: SPECTRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC22_9907-11_SPECTRE; 2024-A02034-43 (Registry Identifier: N° ID-RCB)
Record Dates: First submitted 2024-12-20; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Brain Diseases; Ischemic Stroke; Stroke; Brain Infarction; Stroke Rehabilitation
Keywords: stroke; Rehabilitation; Upper Limb; Neuroplasticity; Connectivity
MeSH Terms: conditions — Brain Diseases; Ischemic Stroke; Stroke; Brain Infarction

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, cohort, interventional study with minimal risks and constraints according to the Loi Jardé (RIPH2).
  Longitudinal follow-up of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Three prognostic groups according to the PREP2 algorithm (good, limited and poor).
  21 evaluable patients divided into 3 balanced prognostic groups.
  Interventions: Other: Clinical scores and functional MRI

INTERVENTIONS:
Other: Clinical scores and functional MRI — Motor evoked potentials between Day 3-Day 7 of the stroke, for a equal distribution of patients into three prognostic groups according to the PREP2 algorithm (good, limited and poor). Longitudinal follow-up with clinical scores and functional MRI at Day 7-Day 10, Day 30, Month 3 and Month 6 of stroke.

SUMMARY:
SPECTRE is a prospective longitudinal study in order to identify whether patients with different degrees of motor recovery are distinguished by distinct brain post-stroke plasticity patterns in the acute and sub-acute phases. This study allows close longitudinal follow-up of patients with severe clinical motor impairment using functional MRI to study cerebral neuroplasticity after ischemic stroke in the acute and sub-acute phase in patients with upper limb motor impairement, taking into account prognostic criteria used in current practice.

DETAILED DESCRIPTION:
Patients are recruited as they are admitted to the neurovascular department. The SAFE score from the Stinear study is taken on Day 3 of the stroke, followed by motor evoked potentials between Day 3-Day 7 of the stroke, for a equal distribution of patients into three prognostic groups according to the PREP2 algorithm (good, limited and poor).

Longitudinal follow-up with clinical scores and functional MRI at Day 7-Day 10, Day 30, Month 3 and Month 6 of stroke.

Patients will ultimately be classified and analyzed according to their effective motor recovery at 6 months, using the Fugl-Meyer score.

The investigators will then conduct a comprehensive analysis of brain connectivity, examining both the anatomical structure of the brain, its functional activity and the dynamic interactions between certain regions of interest over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age greater than or equal to 18 years) less than 75 years of age, both sexes;
* single supratentorial ischemic stroke confirmed by brain imaging
* Upper limb deficit defined by a SAFE score <5 (SAFE Stinear protocol, prognosis of post-stroke upper limb recovery) on D3 of stroke. This corresponds to the sum of shoulder abduction and finger extension according to the MRC (Medical Research Council) scale for each of these movements out of 5.
* Absence of comprehension disorders limiting participation;
* Patient covered by french social security;
* Free, informed and written consent signed by the patient or a member of the patient's family (in the case of a patient who is able to understand the information and give consent but has motor difficulties resulting in an invalid signature).

Non-Inclusion Criteria:

* Multiple ischemic strokes or history of clinically significant stroke ;
* Posterior fossa stroke ;
* Hemorrhagic stroke;
* Patient who have undergone thrombolysis or mechanical thrombectomy;
* Extensive Fazekas grade 3 vascular leukopathy;
* Pre-existing neurodegenerative pathology;
* Patient with severe dyspnea or swallowing disorders who cannot undergo brain MRI;
* Adults under legal protection (safeguard of justice, curatorship, guardianship, family habilitation), persons deprived of liberty;
* Women declaring that they are pregnant or breast-feeding;
* Patient participating in another therapeutic or drug intervention study that may have an impact on the effect of cerebral neuroplasticity on the SPECTRE study;
* Patients with contraindications to MRI pacemaker or implantable defibrillator, neurosurgical clips, cochlear implants, intra-orbital or encephalic metallic foreign bodies, stents placed less than 4 weeks ago and osteosynthesis devices placed less than 6 weeks ago, claustrophobia.

Exclusion Criteria:

* If the prognostic group according to the PREP2 algorithm (good, limited and poor) has already been reached during motor evoked potential assessment the patient is excluded.
* Recurrence of clinically significant stroke (with worsening NIHSS score > 4) during study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in effective connectivity of Brain data (fMRI activity and CST tractography) | 6 months
  Descriptive analysis of topological measures of effective connectivity graphs as a function of effective motor recovery (Fugl-Meyer score - Upper Extremity) at 6 months. The Fugl-Meyer upper limb motor subscale has a maximum score of 66.
  The effective Fugl Meyer score classifies motor recovery into 3 categories (mild, moderate and severe). A Fugl Meyer score of 0-28 is classified as severe, 29-42 as moderate and 42-66 as mild.

SECONDARY OUTCOMES:
Changes in Effective connectivity of brain data | From Day 7-Day 10 to 6 months
  Longitudinal analysis of topological measures of effective connectivity graphs (between Region of interest (ROIs)) according to recovery categories defined by the Fugl-Meyer score.
Changes in Structural connectivity of brain data | From Day7-Day 10 to 6 months
  Analysis of topological measures of structural connectivity graphs according to recovery categories defined by the Fugl-Meyer score.
Changes in Modification of brain activity of brain data | From Day 7-Day 10 to 6 months
  Longitudinal analysis of brain activity (expressed as variation in BOLD hemodynamic response) at rest and during a motor task (between ROIs) according to recovery categories defined by the Fugl-Meyer score.
Changes in Ipsilesional / contralesional laterality index of brain data | From Day 7-Day 10 to 6 months
  Longitudinal analysis of the ipsilesional/counterlesional laterality index of activations in sensorimotor areas according to recovery categories defined by the Fugl-Meyer score.
Changes in perfusion of brain data | From Day 7-Day 10 to 6 months
  Longitudinal analysis of perfusion (infratentorial, interhemispheric, intrahemispheric) according to recovery categories defined by the Fugl-Meyer score.
Changes in Degree of corticospinal FA ratio of brain data | From Day 7-Day 10 to 6 months
  Longitudinal analysis of the degree of FA ratio of the cortico-spinal tract (injured hemisphere / healthy hemisphere) according to the recovery categories defined by the Fugl-Meyer score.
Changes in patients' clinical profile in terms of motricity | 6 months
  Changes in Motor scores Motor index for upper and lower limbs according to recovery categories defined by the Fugl-Meyer score.
  The Motricity Index can be used to assess the motor impairment in a patient who has had a stroke. This test includes a motor test on the upper limb with a score from 0 to 100, combined with a motor test on the lower limb with a score from 0 to 100. The sum of these two scores is divided by 2 for a total out of 100. A high score indicates good recovery."
Changes in patients' clinical profile in terms of motricity | 6 months
  Changes in Action Research Arm Test (ARAT) score according to recovery categories defined by the Fugl-Meyer score.
  The total score on the ARAT ranges from 0 to 57, with the lowest score indicating that no movements can be performed, and the upper score indicating normal performance. Thus, higher scores will indicate better performance. The ARAT scores is a continuous measure, with no categorical cutoff scores.
Changes in patients' clinical profile in quality of life | 6 months
  Progression in The Stroke Impact Scale (SIS) score according to recovery categories defined by the Fugl-Meyer score.
  The SIS contains 59 items measuring eight domains: strength (4 items), hand functionality (5 items), ADL / IADL (10 items), mobility (9 items), communication (7 items), emotions (9 items), memory / thinking (7 items), and social participation (8 items). A final item assessing overall stroke recovery is asked of the patient (score out of 100).
  The minimum score is 60, the maximum is 300. A high score indicates a good quality of life.
Changes in patients' clinical profile in independence | 6 months
  Progression in The Composite Functional Independence Scale (MIF) score according to recovery categories defined by the Fugl-Meyer score.
  The MIF consists of 18 items measuring patients' performance in performance in activities of daily living, including cognitive and relational aspects. For each item (from 1 to 18), the therapist chooses the patient's level of incapacity from 1 (total assistance) to 7 (total independence). The total score is calculated by adding up the disability level figures for each item. The minimum score is 18, the maximum is 126. A high score indicates complete independence.
Changes in patients' clinical profile in spasticity | 6 months
  Progression in Changes in Tardieu Scale according to recovery categories defined by the Fugl-Meyer score.
  The Tardieu Scale are clinical measures of muscle spasticity in patients with neurological conditions. The Tardieu Scale quantify spasticity by assessing the muscle's response to stretch applied at given velocities. The examiner evaluates the muscle group's reaction to stretch at a specified velocity with 2 parameters: X (quality of muscle reaction) and Y (angle of muscle reaction).
Changes in clinical profile in terms of motor skills | Day 7-Day 10
  Changes in Fugl-Meyer Assesment - Upper Extremity (FMA-UE) according to recovery categories defined by the Fugl-Meyer score.
  The FMA assesses motor impairment of the upper and lower limb, balance, sensitivity, passive joint mobility and pain on mobilization following stroke.
  The Fugl-Meyer upper limb motor subscale has a maximum score of 66. The effective Fugl Meyer score classifies motor recovery into 3 categories (mild, moderate and severe). A Fugl Meyer score of 0-28 is classified as severe, 29-42 as moderate and 42-66 as mild.
Changes in clinical profile in terms of motor skills | Day 30
  Changes in Fugl-Meyer Assesment - Upper Extremity (FMA-UE) according to recovery categories defined by the Fugl-Meyer score.
  The FMA assesses motor impairment of the upper and lower limb, balance, sensitivity, passive joint mobility and pain on mobilization following stroke.
  The Fugl-Meyer upper limb motor subscale has a maximum score of 66. The effective Fugl Meyer score classifies motor recovery into 3 categories (mild, moderate and severe). A Fugl Meyer score of 0-28 is classified as severe, 29-42 as moderate and 42-66 as mild.
Changes in clinical profile in terms of motor skills | 3 months
  Changes in Fugl-Meyer Assesment - Upper Extremity (FMA-UE) according to recovery categories defined by the Fugl-Meyer score.
  The FMA assesses motor impairment of the upper and lower limb, balance, sensitivity, passive joint mobility and pain on mobilization following stroke.
  The Fugl-Meyer upper limb motor subscale has a maximum score of 66. The effective Fugl Meyer score classifies motor recovery into 3 categories (mild, moderate and severe). A Fugl Meyer score of 0-28 is classified as severe, 29-42 as moderate and 42-66 as mild.
Changes in clinical profile in terms of motor skills | 6 months
  Changes in Fugl-Meyer Assesment - Upper Extremity (FMA-UE) according to recovery categories defined by the Fugl-Meyer score.
  The FMA assesses motor impairment of the upper and lower limb, balance, sensitivity, passive joint mobility and pain on mobilization following stroke.
  The Fugl-Meyer upper limb motor subscale has a maximum score of 66. The effective Fugl Meyer score classifies motor recovery into 3 categories (mild, moderate and severe). A Fugl Meyer score of 0-28 is classified as severe, 29-42 as moderate and 42-66 as mild.
Changes in clinical profile in terms of of global impairment | Day 7-Day 10
  Changes in National Institutes of Health Stroke Scale (NIHSS) according to recovery categories defined by the Fugl-Meyer score.
  This scale assesses level of consciousness, extraocular movements, field of vision, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria) and hemineglect (neglect). Total NIHSS scores range from 0 to 42, with higher values reflecting more severe brain damage. Stroke severity is defined according to threshold scores as follows: > 25 - severe neurological deficits, 5-14 - moderate neurological deficits, < 5 - mild deficits.
Changes in clinical profile in terms of of global impairment | Day 30
  Changes in National Institutes of Health Stroke Scale (NIHSS) according to recovery categories defined by the Fugl-Meyer score.
  This scale assesses level of consciousness, extraocular movements, field of vision, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria) and hemineglect (neglect). Total NIHSS scores range from 0 to 42, with higher values reflecting more severe brain damage. Stroke severity is defined according to threshold scores as follows: > 25 - severe neurological deficits, 5-14 - moderate neurological deficits, < 5 - mild deficits.
Changes in clinical profile in terms of of global impairment | 3 months
  Changes in National Institutes of Health Stroke Scale (NIHSS) according to recovery categories defined by the Fugl-Meyer score.
  This scale assesses level of consciousness, extraocular movements, field of vision, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria) and hemineglect (neglect). Total NIHSS scores range from 0 to 42, with higher values reflecting more severe brain damage. Stroke severity is defined according to threshold scores as follows: > 25 - severe neurological deficits, 5-14 - moderate neurological deficits, < 5 - mild deficits.
Changes in clinical profile in terms of of global impairment | 6 months
  Changes in National Institutes of Health Stroke Scale (NIHSS) according to recovery categories defined by the Fugl-Meyer score.
  This scale assesses level of consciousness, extraocular movements, field of vision, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria) and hemineglect (neglect). Total NIHSS scores range from 0 to 42, with higher values reflecting more severe brain damage. Stroke severity is defined according to threshold scores as follows: > 25 - severe neurological deficits, 5-14 - moderate neurological deficits, < 5 - mild deficits.
Changes in neurological events | From enrollment to the end of evaluation at 6 months
  Changes in significant clinical worsening defined by a worsening of the NIHSS score by 4 points, epileptic seizure.
  This scale assesses level of consciousness, extraocular movements, field of vision, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria) and hemineglect (neglect). Total NIHSS scores range from 0 to 42, with higher values reflecting more severe brain damage. Stroke severity is defined according to threshold scores as follows: > 25 - severe neurological deficits, 5-14 - moderate neurological deficits, < 5 - mild deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Maud GUILLEN, Md, Principal Investigator — RENNES CHU
Locations (1):
- Rennes Chu, Rennes, France, France

IPD SHARING:
Plan to Share IPD: Undecided